CLINICAL TRIAL: NCT03611023
Title: Multicentric Observational Study of the Touch® Trapezo-metacarpal Prosthesis
Brief Title: Study of the Touch® Trapezo-metacarpal Prosthesis
Status: Active, not recruiting | Type: Observational
Sponsor: Groupe Concepteur Touch (Other)
Responsible Party: Principal Investigator, Dr Cyril Falaise, Principal Investigator, Groupe Concepteur Touch
Other Study IDs: 2018-01
Record Dates: First submitted 2018-07-09; First posted 2018-08-02 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Complications Due to Internal Joint Prosthesis; Thumb Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational study of implanted patients with a new orthopaedic implant: the Touch trapezo-metacarpal prosthesis

DETAILED DESCRIPTION:
Prospective observational study of implanted patients with a new orthopaedic implant: the Touch double mobility trapezo-metacarpal prosthesis, 15 years follow up.

ELIGIBILITY:
Inclusion Criteria:

• Patients implanted with the Touch® prosthesis by one of the three investigating surgeons

Exclusion Criteria:

* Patient not in capacity to understand the study
* Patient not in capacity to consent to the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with the Touch® prosthesis by one of the three investigating surgeons
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2036-09 (Estimated); Study Completion 2036-09 (Estimated)

PRIMARY OUTCOMES:
Implant Survival at 3 years | 3 Years
  Failure rate of the implant
Implant Survival at 5 years | 5 Years
  Failure rate of the implant
Implant Survival at 10 years | 10 Years
  Failure rate of the implant
Implant Survival at 15 years | 15 Years
  Failure rate of the implant

SECONDARY OUTCOMES:
Functional Outcome at 3 years | 3 Years
  QuickDASH score (Disabilities of the Arm, Shoulder and Hand score, is the mean result of 11 questions regarding patient ability to perform everyday activities), 0 to 100, with 0 the better
Functional Outcome at 5 years | 5 Years
  QuickDASH score (Disabilities of the Arm, Shoulder and Hand score, is the mean result of 11 questions regarding patient ability to perform everyday activities), 0 to 100, with 0 the better
Functional Outcome at 10 years | 10 Years
  QuickDASH score (Disabilities of the Arm, Shoulder and Hand score, is the mean result of 11 questions regarding patient ability to perform everyday activities), 0 to 100, with 0 the better
Functional Outcome at 15 years | 15 Years
  QuickDASH score (Disabilities of the Arm, Shoulder and Hand score, is the mean result of 11 questions regarding patient ability to perform everyday activities), 0 to 100, with 0 the better

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital du Gier, Saint-Chamond, France

IPD SHARING:
Plan to Share IPD: No